CLINICAL TRIAL: NCT01248442
Title: Placebo Controlled Study to Assess the Effects of Vitamin D Supplementation on Parameters of the Immune, Endocrine and Metabolic System in Healthy Women and Men.
Brief Title: Immune and Metabolic Effects of Vitamin D Supplementation in Healthy Humans
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ENM-EA-011
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Healthy Humans
Keywords: Vitamin D Deficiency; Autoimmune disease; Diabetes
MeSH Terms: conditions — Vitamin D Deficiency; Autoimmune Diseases; Diabetes Mellitus | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cholecalciferol (Experimental)
  Interventions: Drug: Cholecalciferol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cholecalciferol — monthly dose of 140.000 IU of cholecalciferol orally, 3 times.
  Other Names: Oleovit D3
  Arms: Cholecalciferol
Drug: Placebo — Matching Placebo
  Other Names: Almondoil
  Arms: Placebo

SUMMARY:
In this placebo controlled study the investigators aim to investigate the effect of a 3 month vitamin D supplementation on parameters of the immune, endocrine and metabolic system in healthy women and men. Vitamin D. In a pilot study the investigators showed an increase of certain immune cells, which regulate immunotolerance, the investigators therefore try to confirm these results with a placebo group. Furthermore the investigators assess the effect of vitamin D on the glucose metabolism and hormone levels.

DETAILED DESCRIPTION:
This is a randomized double-blind placebo controlled trial, with the aim to investigate the effect of a Vitamin D supplementation on parameters of the immune, endocrine and metabolic system in healthy humans without diabetes and obesity.

The primary aim is to assess the effect of vitamin D supplementation of the number and function of peripheral regulatory T-cells (Tregs). The investigators will measure the Tregs at baseline and monthly for 3 months. Furthermore the investigators assess additional immune cells from the adaptive immunosystem.

Furthermore the investigators will perform a standard mixed meal tolerance test at baseline and 3 months following the supplementation in order to assess the insulin secretion in vivo.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 10 years
* healthy subjects without chronic disease

Exclusion Criteria:

* Hypercalcemia >2,65 mmol/L
* pregnancy and lactation period
* acute infections
* chronic disease requiring treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Increase and function of peripheral regulatory T-cells | 3 months
  The level and function of the regulatory T-cells will be compared between the two groups.

SECONDARY OUTCOMES:
immunophenotyping | 3 months
  The effect of vitamin D on circulating immune cells and cytokine secretion will be measured at basal and after 3 months.
Renin and aldosterone concentrations | 3 months
  serum renin and aldosterone levels will be measured basal and after 3 months.
Insulin secretion | 3 months
  Insulin secretion assessed with a mixed meal tolerance test will be performed basal and after 3 months
calcium levels | 3 months
  serum calcium levels will be measured basal and monthly for 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Pieber, Prof., Principal Investigator — Medical University of Graz
Locations (1):
- Medical University Graz, Graz, Austria

REFERENCES:
- [Derived] Prietl B, Treiber G, Mader JK, Hoeller E, Wolf M, Pilz S, Graninger WB, Obermayer-Pietsch BM, Pieber TR. High-dose cholecalciferol supplementation significantly increases peripheral CD4(+) Tregs in healthy adults without negatively affecting the frequency of other immune cells. Eur J Nutr. 2014 Apr;53(3):751-9. doi: 10.1007/s00394-013-0579-6. Epub 2013 Sep 3. PMID 23999998